CLINICAL TRIAL: NCT00695071
Title: Assessment of the Steady State Pharmacokinetics of Itraconazole and Hydroxy-Itraconazole in Healthy Subjects After Administration of a New Itraconazole 200 mg Film Coated Tablet Once Daily for Fourteen Days in Fed Condition
Brief Title: Study to Assess Blood Levels of Itraconazole During a Two-Week Period
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: BT0300-108-USA
Record Dates: First submitted 2008-06-09; First posted 2008-06-11 (Estimated); Last update posted 2011-09-26 (Estimated); Status verified 2011-09

CONDITIONS: Healthy
Keywords: Healthy Volunteers
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Active Comparator)
  Interventions: Drug: Itraconazole

INTERVENTIONS:
Drug: Itraconazole — Oral

SUMMARY:
The objective of this clinical trial is to document the steady state pharmacokinetics and safety of a new itraconazole 200 mg film coated tablet.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.0 and 28.0 kg/m2
* Good physical and mental health status, determined on the basis of the medical history and a general clinical examination.
* Vital signs (blood pressure and heart rate) in supine position within the normal range
* Electrocardiogram (12 lead) considered as normal
* Non-smoker.
* Able to swallow pills
* If subject is a woman of childbearing potential (WOCBP), must agree to use adequate birth control as defined by the protocol

Exclusion Criteria:

* Any disease or physical condition which, in the opinion of the investigator, could impact the pharmacokinetics of the drug
* History or presence of drug abuse or consumption of alcohol
* History of sensitivity or allergy to azoles or related drugs
* Any requirement to be on other drug treatment (except acetaminophen and for WOCBP, hormonal contraceptives)
* Unsuitable veins for repeated venipuncture.
* Clinically significant abnormal ECG
* Nursing mothers and pregnant women, or women of childbearing potential not using adequate contraceptives.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2008-06; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Steady State Plasma levels of Itraconazole | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (1):
- Advanced Biomedical Research, Hackensack, New Jersey, United States